CLINICAL TRIAL: NCT06376630
Title: Study of Microvascular Dysfunction, Coronary Flow Reserve and Cardioprotective Effect of Early Intravenously Administration of Esmolol in Patients With Myocardial Infarction
Brief Title: Study of Microvascular Dysfunction, CFR and Cardioprotective Effect of Early Administration of Esmolol in MI
Acronym: ESMO-VASCMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Principal Investigator, Dmitry Pevzner, Head of the Emergency Cardiology Department, National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 298-2024
Record Dates: First submitted 2024-04-10; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Myocardial Infarction; Coronary Stenosis; Coronary Microvascular Dysfunction
MeSH Terms: conditions — Myocardial Infarction; Coronary Stenosis | interventions — esmolol

STUDY DESIGN:
Intervention Model Description: 300 pts with MI are to be enrolled. Among them 100 pts with STEMI will be included into the substudy evaluating cardioprotective effects of early iv administration of esmolol. They will be randomized 1:1 by in arms receiving esmolol or no IV beta-blockers. In the esmolol arm the infusion will begin immediately on admission. 200 pts with MI and multivessel disease with non-IRA lesions of 50-85% diameter stenosis will be included into another substudy investigating coronary physiology. All patients will undergo PCI with IRA stenting. 50 stable patients will undergo invasive measurements of coronary physiology. Those will also undergo cardiac MRI. Other 150 pts will not undergo invasive measurements of coronary physiology during initial hospitalization. Pts in both groups will be hospitalized again in 30-40 days after MI. They will undergo stress SPECT or stress echocardiography. All patients will undergo a follow-up coronary angiography with invasive measurement of coronary physiology.
Who Masked: Investigator
Masking Description: envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Substudy evaluating cardioprotective effects of early iv administration of esmolol (Active Comparator): 100 pts with STEMI will be randomized 1:1 in arms receiving esmolol or no IV beta-blockers. In the esmolol arm the infusion will begin immediately on admission
  Interventions: Drug: Esmolol Hcl 10Mg/Ml Inj
- Substudy investigating coronary physiology (No Intervention): 50 stable patients with MI will undergo invasive measurements of coronary physiology. Those will also undergo cardiac MRI. Other 150 pts will not undergo invasive measurements of coronary physiology during initial hospitalization. Pts in both groups will be hospitalized again in 30-40 days after MI. They will undergo stress SPECT or stress echocardiography. All patients will undergo a follow-up coronary angiography with invasive measurement of coronary physiology

INTERVENTIONS:
Drug: Esmolol Hcl 10Mg/Ml Inj — the loading dose of 500 mkg/kg for 1 minute, followed by the initial rate of 50 mkg/kg/min. Individual titration depending on the desired hemodynamical effect (to the heart rate of 60 bpm or to the maximum tolerated dose maintaining stable hemodynamics) every 5-15 minutes (the maximum allowed rate of administration is 300 mkg/kg/min) for 6 hours.
  Thereafter patients in both treatment arms - the IV esmolol arm and the placebo arm, will be administered oral β-adrenergic blockers, if decided so by the treating physician and unless contraindicated.
  Other Names: Esmolol
  Arms: Substudy evaluating cardioprotective effects of early iv administration of esmolol

SUMMARY:
Study rationale: to evaluate clinical and prognostic relevance of microvascular dysfunction, coronary flow reserve and cardioprotective effects of iv administration of esmolol in patients with myocardial infarction.

First substudy is an open randomized trial evaluating the efficacy and safety of early intravenous administration of esmolol in patients with acute ST-segment elevation myocardial infarction (MI) and relative contraindications to administration of other intravenous β1-adrenergic blocker (metoprolol etс.). Сomparison group will include patients who have not received intravenous β1-adrenergic blocker. Secondary outcome in this substudy is the degree of microvascular obstruction and infarct size according to MRI with gadolinium delayed enhancement.

Second substudy examines the quantitative parameters of coronary physiology in patients with MI and multivessel disease. Changes of coronary physiology measurements over time ((iFR, Pd/Pa, FFR, delta FFR, gradient FFR per time unit (dFFR(t)/dt), pullback pressure gradient (PPG)) measured in the infarct-related artery and in non-infarct-related arteries with diameter stenosis of 50-85% immediately after the completion of a primary percutaneous coronary intervention and during a second hospitalization (30-45 days after STEMI) will be evaluated. The comparison changes of coronary physiology over time with presence of an MVO and infarct size determined by MRI. The model of calculating coronary flow reserve (CFR) based on tridimensional reconstruction of coronary arteries and coronary physiology parameters as measured during coronary angiography will be developed. The influence of coronary physiology parameters measured after complete myocardial revascularization by PCI, and derived CFR in patients with MI on long-term clinical outcomes will be evaluated, based on prospective data collection.

Primary composite outcome in all substudies will be the sum of adverse cardiac outcomes (congestive heart failure, episodes of recurrent congestive heart failure worsening resulting in hospitalizations, cardiac mortality, MI recurrences, unstable angina, urgent myocardial revascularization) within > 12 months post-infarction.

Secondary composite outcome in all substudies is the degree of microvascular obstruction and infarct size evaluated by MRI with gadolinium delayed enhancement.

DETAILED DESCRIPTION:
Study rationale: to evaluate clinical and prognostic relevance of microvascular dysfunction, coronary flow reserve and cardioprotective effects of iv administration of esmolol in patients with myocardial infarction.

Substudy of early esmolol administration: On admission patients will undergo ECG and echocardiography in an intensive care ward, according to standard clinical practice. Eligible patients having signed the Informed Consent Form will be randomized 1:1 by appropriate software. In the esmolol arm the infusion will begin immediately on admission simultaneously with conventional upfront treatment. Study procedures will be performed in parallel to the patient's preparation for the catheterization lab and transportation for primary PCI, without any delay of time to the catheterization lab. During the hospitalization cardiac MRI will be done with contrast enhancement using an ultraconducting MRI scanner with the magnetic field intensity of 1.5 T (Siemens Avanto). The following elements will be done without contrast enhancement:

* cine imaging MRI in standard views (long axis 2- and 4-chamber views, LV short axis) measuring left ventricle end diastolic volume (LV EDV), left ventricle end systolic volume (LV ESV), LV EF, regional wall motion abnormality across 17 LV segments;
* Т2-weighed images (T2WI) using the same views to assess myocardial edema (signal intensity elevation more than 2-fold compared to the normal myocardium).

For contrast enhancement a gadolinium-based contrast agent will be used (gadobutrol, Bayer) in the dose of 0.15 mmol/kg body weight. The following elements will be done with contrast enhancement:

* early contrast enhancement (2 minutes after intravenous administration of the contrast agent);
* delayed contrast enhancement (10 - 20 minutes after intravenous administration of the contrast agent).

The areas demonstrating with contrast enhancement will be assessed as areas of acute or chronic myocardial injury (during the presence of edema, according to T2WI results).

Substudy investigating coronary physiology. This substudy is expected to include 200 patients with MI and multivessel Coronary Artery Disease who will be found on PCI (performed for the IRA) to have lesions with diameter stenosis of 50-85% in other arteries.

During hospitalization for AMI treatment and diagnostic evaluation of patients will be done according to current clinical practice guidelines. All patients enrolled into the study will undergo PCI with IRA stenting. In the STEMI group, 50 hemodynamically stable patients after primary PCI will undergo invasive measurements of coronary hemodynamical parameters: instantaneous wave-free ratio, Pd/Pa, FFR with papaverine administration both into the IRA and into non-IRA (FFR measurements with papaverine administration will only be performed in patients without contraindications to such administrations [as worded for AMI patients as a separate exclusion criterion]). During the hospitalization those 50 patients will undergo cardiac MRI with IV contrast enhancement to evaluate MVO, beyond routine assessments.

Other 150 patients enrolled into the study (50 with STEMI and 100 with NSTEMI) during their first hospitalization for AMI will only undergo routine assessments and treatment procedures according to clinical practice guidelines. In 30-40 days after the MI patients will be hospitalized again. During their second hospitalization patients will undergo stress SPECT myocardial perfusion imaging or exercise stress echocardiography with physical exertion or ATP infusion, with CFR measurement, unless contraindicated. All patients will undergo a follow-up coronary angiography with invasive measurement of coronary hemodynamical parameters in non-IRA, accompanied by an assessment of IRA stenting outcomes (instantaneous wave-free ratio, Pd/Pa, unless contraindicated - FFR with papaverine administration etc.). If non-IRA stenting is indicated, PCI with subsequent invasive re-assessment of coronary hemodynamical parameters. The CFR value across the coronary artery basins will be calculated based on the tridimensional reconstruction of coronary arteries and intracoronary pressure measurements before and after stenting. In the subgroup of patients who underwent measurements of coronary hemodynamical parameters in the acute setting, follow-up measurements of coronary hemodynamical parameters will be performed. Subsequently relationship will be evaluated between invasive measurements of coronary hemodynamical parameters and the presence of MVO. Also, results of stress tests will be compared to invasive measurements of coronary hemodynamical parameters. Patients demonstrating CFR reduction in a stress echocardiography with ATP infusion will be asked to repeat a stress test within 1 month post-stenting, during a hospitalization, or on an out-patient visit within one month after discharge from the hospital.

ELIGIBILITY:
Substudy evaluating cardioprotective effects of early iv administration of esmolol

Inclusion Criteria:

* Diagnosed acute ST elevation MI, type 1, within the first 8 hours of disease onset;
* Treating physician's decision not to administer metoprolol intravenously prior to primary PCI due to a high risk of complications (BP < 120/80 mm Hg at baseline examination, moderate evidence of heart failure (Killip 2) or a risk of its development (LV EF ≤ 30%), first degree AV block with PQ ≥ 0.25 ms, history of asthma or severe COPD etc.)
* Signed Informed Consent to participate in the study

Exclusion Criteria:

* severe heart failure (pulmonary edema; SCAI В-Е cardiogenic shock);
* atrioventricular conduction abnormality higher than first degree, without a pacemaker;
* sinus bradycardia with the heart rate of < 60 bpm;
* BP < 100/60 mm Hg.;
* asthma in exacerbation;
* history of a STEMI in the IRA basin;
* clinically significant bleeding or hypovolemia;
* hypersensitivity to esmolol;
* pregnancy or lactation;
* known severe comorbidities independently affecting prognosis (Child Pugh class C liver failure, active malignancies etc.);
* contraindications to MRI (MR-incompatible pacemaker/implanted cardioverter-defibrillator, cochlear implants, clips on brain vessels, foreign metal objects - bullets, intraorbital metal fragments, insulin pumps, body weight above 150 kg, history of allergies to gadolinium, claustrophobia);
* severe dementia;
* known severe comorbidities independently affecting prognosis (chronic renal or liver failure, active malignancies etc.);
* complicated PCI, "no reflow" phenomenon on follow-up coronary angiography;
* thrombolysis for AMI;
* ECG evidence of spontaneous reperfusion on admission;
* patient's refusal from participation in the study.

Substudy investigating coronary physiology

Inclusion Criteria:

* Diagnosed MI, completed PCI for the IRA and multivessel Coronary Artery Disease with diameter stenosis of 50-85% in non-IRA.
* Signed Informed Consent to participate in the study

Exclusion criteria:

* History of coronary artery bypass grafting surgery;
* Non-IRA lesions resulting in diameter stenosis of below 50% and above 85%, main left coronary artery (LCA) stenosis above 50%;
* Chronic kidney disease stage 3b or above (glomerular filtration rate below 45 mL/min/m2 according to the CKD-EPI equation);
* History of a contrast-induced nephropathy (CIN) or a high CIN risk (calculated using the Mehran score);
* History of allergies to iodine-containing medications;
* Pregnancy or lactation;
* Left ventricle ejection fraction ≤ 30%;
* Known severe comorbidities independently affecting prognosis (chronic renal or liver failure, active malignancies etc.);
* Early post-infarction angina;
* Severe dementia;
* Patient's refusal from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2029-01-29 (Estimated); Study Completion 2030-01-29 (Estimated)

PRIMARY OUTCOMES:
Composite of adverse cardiac outcomes | Through study completion, an average of 2 years
  Congestive heart failure, episodes of recurrent congestive heart failure worsening resulting in hospitalizations, cardiac mortality, MI recurrences, unstable angina, urgent myocardial revascularization

SECONDARY OUTCOMES:
Degree of microvascular obstruction | During the week after myocardial infarction
  Evaluation by MRI with gadolinium delayed enhancement
Infarct size | During the week after myocardial infarction
  Evaluation by MRI with gadolinium delayed enhancement

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Pevzner, MD, Principal Investigator — National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Locations (1):
- NMRCCardiologyRu, Moscow, Russia

REFERENCES:
- [Background] Sun B, Wang CY, Chen RR. Clinical Efficacy and Safety of Early Intravenous Administration of Beta-Blockers in Patients Suffering from Acute ST-Segment Elevation Myocardial Infarction Without Heart Failure Undergoing Primary Percutaneous Coronary Intervention: A Study-Level Meta-Analysis of Randomized Clinical Trials. Cardiovasc Drugs Ther. 2024 Aug;38(4):833-846. doi: 10.1007/s10557-023-07448-x. Epub 2023 Apr 1. PMID 37002468
- [Background] Garcia-Ruiz JM, Fernandez-Jimenez R, Garcia-Alvarez A, Pizarro G, Galan-Arriola C, Fernandez-Friera L, Mateos A, Nuno-Ayala M, Aguero J, Sanchez-Gonzalez J, Garcia-Prieto J, Lopez-Melgar B, Martinez-Tenorio P, Lopez-Martin GJ, Macias A, Perez-Asenjo B, Cabrera JA, Fernandez-Ortiz A, Fuster V, Ibanez B. Impact of the Timing of Metoprolol Administration During STEMI on Infarct Size and Ventricular Function. J Am Coll Cardiol. 2016 May 10;67(18):2093-2104. doi: 10.1016/j.jacc.2016.02.050. Epub 2016 Apr 3. PMID 27052688
- [Background] Er F, Dahlem KM, Nia AM, Erdmann E, Waltenberger J, Hellmich M, Kuhr K, Le MT, Herrfurth T, Taghiyev Z, Biesenbach E, Yuksel D, Eran-Ergoknil A, Vanezi M, Caglayan E, Gassanov N. Randomized Control of Sympathetic Drive With Continuous Intravenous Esmolol in Patients With Acute ST-Segment Elevation Myocardial Infarction: The BEtA-Blocker Therapy in Acute Myocardial Infarction (BEAT-AMI) Trial. JACC Cardiovasc Interv. 2016 Feb 8;9(3):231-240. doi: 10.1016/j.jcin.2015.10.035. PMID 26847114
- [Background] Clemente-Moragon A, Gomez M, Villena-Gutierrez R, Lalama DV, Garcia-Prieto J, Martinez F, Sanchez-Cabo F, Fuster V, Oliver E, Ibanez B. Metoprolol exerts a non-class effect against ischaemia-reperfusion injury by abrogating exacerbated inflammation. Eur Heart J. 2020 Dec 7;41(46):4425-4440. doi: 10.1093/eurheartj/ehaa733. PMID 33026079
- [Background] Van Herck PL, Paelinck BP, Haine SE, Claeys MJ, Miljoen H, Bosmans JM, Parizel PM, Vrints CJ. Impaired coronary flow reserve after a recent myocardial infarction: correlation with infarct size and extent of microvascular obstruction. Int J Cardiol. 2013 Jul 31;167(2):351-6. doi: 10.1016/j.ijcard.2011.12.099. Epub 2012 Jan 13. PMID 22244483
- [Background] Anderson HVS. Acute Coronary Physiology. JACC Cardiovasc Interv. 2020 May 25;13(10):1168-1170. doi: 10.1016/j.jcin.2020.03.037. No abstract available. PMID 32438987
- [Background] Kelshiker MA, Seligman H, Howard JP, Rahman H, Foley M, Nowbar AN, Rajkumar CA, Shun-Shin MJ, Ahmad Y, Sen S, Al-Lamee R, Petraco R; Coronary Flow Outcomes Reviewing Committee. Coronary flow reserve and cardiovascular outcomes: a systematic review and meta-analysis. Eur Heart J. 2022 Apr 19;43(16):1582-1593. doi: 10.1093/eurheartj/ehab775. PMID 34849697
- [Background] Lee JM, Lee SH, Shin D, Choi KH, van de Hoef TP, Kim HK, Samady H, Kakuta T, Matsuo H, Koo BK, Fearon WF, Escaned J. Physiology-Based Revascularization: A New Approach to Plan and Optimize Percutaneous Coronary Intervention. JACC Asia. 2021 May 21;1(1):14-36. doi: 10.1016/j.jacasi.2021.03.002. eCollection 2021 Jun. PMID 36338358
- [Background] Hausenloy DJ, Chilian W, Crea F, Davidson SM, Ferdinandy P, Garcia-Dorado D, van Royen N, Schulz R, Heusch G. The coronary circulation in acute myocardial ischaemia/reperfusion injury: a target for cardioprotection. Cardiovasc Res. 2019 Jun 1;115(7):1143-1155. doi: 10.1093/cvr/cvy286. PMID 30428011
- [Background] Csippa B, Uveges A, Gyurki D, Jenei C, Tar B, Bugarin-Horvath B, Szabo GT, Komocsi A, Paal G, Koszegi Z. Simplified coronary flow reserve calculations based on three-dimensional coronary reconstruction and intracoronary pressure data. Cardiol J. 2023;30(4):516-525. doi: 10.5603/CJ.a2021.0117. Epub 2021 Oct 8. PMID 34622434
- [Background] Terenicheva MA, Shakhnovich RM, Stukalova OV, Pevzner DV, Arutyunyan GK, Demchenkova AY, Merkulova IN, Ternovoy SK. Correlations between clinical and laboratory findings and prognostically unfavorable CMR-based characteristics of acute ST-elevation myocardial infarction. Kardiologiia. 2021 Feb 10;61(1):44-51. doi: 10.18087/cardio.2021.1.n1373. English, Russian. PMID 33734055
- [Background] Terenicheva MA, Stukalova OV, Shakhnovich RM, Ternovoy SK. [The role of cardiac magnetic resonance imaging (cardiovascular magnetic resonance) in defining the prognosis of patients with acute ST-segment elevation myocardial infarction. Part 1. Indications and contraindications to cardiovascular magnetic resonance]. Ter Arkh. 2021 Apr 15;93(4):497-501. doi: 10.26442/00403660.2021.04.200687. Russian. PMID 36286787
- [Background] Terenicheva MA, Stukalova OV, Shakhnovich RM, Ternovoy SK. [The role of cardiac magnetic resonance imaging in defining the prognosis of patients with acute ST-segment elevation myocardial infarction. Part 2. Assessment of the disease prognosis]. Ter Arkh. 2022 May 26;94(4):552-557. doi: 10.26442/00403660.2022.04.201458. Russian. PMID 36286807